CLINICAL TRIAL: NCT05354596
Title: Stereotactic Radiation Therapy In Centrally Located Lung and Ultra-centrally Located Tumors in the Lung. STRICT-LUNG & STAR-LUNG STUDY
Brief Title: A Multicenter Phase II Study of Stereotactic Radiotherapy for Centrally Located Lung Tumors (STRICT-LUNG STUDY) and Ultra-centrally Located Lung Tumors (STAR-LUNG STUDY).
Acronym: STRICTSTARLUNG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Odense University Hospital (Other); Vejle Hospital (Other); University of Copenhagen (Other); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Mette Pøhl, MD PhD, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-21041667
Record Dates: First submitted 2022-04-18; First posted 2022-04-29 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer; Metastases to Lung; Radiotherapy Side Effect
Keywords: Stereotactic body radiotherapy (SBRT)
MeSH Terms: conditions — Lung Neoplasms; Radiation Injuries | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Radiation: SBRT of central located and ultra-centrally located tumors in the lung. Primary lung tumors and lung metastasis from solid tumors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STRICT LUNG (Experimental): Central Tumors in the Lung The tumor is considered central when the tumor is located within 0.5 -2.5 cm in all directions of the PBT or the esophagus. The PBT includes trachea, main bronchi and intermediate bronchus and 5 lobar bronchi. In addition, the tumor is also considered central, if it is located <0.5 cm from the spinal cord, heart and aorta.
  Interventions: Procedure: STRICT LUNG
- STAR LUNG (Experimental): Ultra-Centrally Tumors in the Lung Ultra-centrally located tumors are tumors located within the 0.0 to 0.5 cm zone of trachea, main bronchi or intermediate bronchus. The patient will be excluded if the tumor invades the trachea, bronchi, esophagus, or pericardium/heart (radiological or by bronchoscopy assessment).
  Interventions: Procedure: STAR LUNG

INTERVENTIONS:
Procedure: STRICT LUNG — Stereotactic body radiation therapy: Centrally located tumors are treated on standard-linacs with daily CBCT image-guidance and plan adaptation.
  Other Names: Stereotactic radiotherapy for centrally located lung tumors
  Arms: STRICT LUNG
Procedure: STAR LUNG — Stereotactic body radiation therapy: Ultra-centrally tumors are treated on MR-linacs with daily MR-guided plan-adaptation.
  Other Names: Stereotactic radiotherapy for ultra-centrally located lung tumors
  Arms: STAR LUNG

SUMMARY:
An open-label phase II study, investigating toxicity, treatment efficacy and the local tumor control rate in 69 patients with centrally located tumors and in 69 patients with ultra-centrally located tumors in the lung. Treatment and patient outcomes will be recorded. Centrally located tumors are treated on standard-linacs with daily CBCT image-guidance and plan adaptation. Ultra-centrally tumors are treated on MR-linacs with daily MR-guided plan-adaptation.

DETAILED DESCRIPTION:
The STRICT-LUNG study will evaluate the feasibility and safety of daily image-guided SBRT in centrally located lung tumors (primary, oligo-metastatic or oligo-progressive). The STAR-LUNG study will evaluate the feasibility and safety of daily adaptive MR-linac based SBRT in ultra-centrally located lung tumors (primary, oligo-metastatic or oligo-progressive).

The tumor is considered central when the tumor is located within 0.5 -2.5 cm in all directions of the PBT or the esophagus. The PBT includes trachea, main bronchi and intermediate bronchus and 5 lobar bronchi. In addition, the tumor is also considered central, if it is located <0.5 cm from the spinal cord, heart and aorta.

Ultra-centrally located tumors are tumors located within the 0.0 to 0.5 cm zone of trachea, main bronchi or intermediate bronchus. The patient will be excluded if the tumor invades the trachea, bronchi, esophagus, or pericardium/heart (radiological or by bronchoscopy assessment).

The main purposes are to evaluate the feasibility, safety and efficacy of stereotactic radiation to centrally and ultra-centrally located tumors, including treatment related adverse events, quality of life (QoL) assessments, local tumor control rate, disease free survival, and overall survival and facilitate future stratification of this patient group for definitive treatment.

Treatment related adverse events (TRAE) will be registered at baseline, end of treatment, 4-6 weeks, 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, 54, 60 months after treatment, and hereafter every year until 10th year of follow-up.

Enrolment in both trial categories may continue until the required numbers in both groups have been reached.

ELIGIBILITY:
Inclusion Criteria:

* Histology or cytology proven non-hematological cancer or known cancer with local progressive recurrence.
* ECOG performance status ≤ 2.
* Age > 18 years old. • Life expectancy > 6 months.
* Maximum one central tumor with the diameter ≤ 5 cm or > 1 adjacent located tumors with a summarized diameter (measured from the outer margin from one tumor to the outer margin of the other) of maximum 5 cm on a diagnostic CT-scan.
* Medically inoperable or refused surgery.
* The central tumors must be localized within or touching the 2.5 cm-zone of the PBT, or within 0.5 cm from the spinal cord, esophagus or heart. Evaluation is primarily performed on the diagnostic CT scan
* All metastatic sites are treated or planned for ablative therapy (including surgery). For oligo-progressive disease (OPD), only the sites in progression are required to fulfil this criterion
* Adequate lung function to tolerate treatment, at the discretion of the treating physician. • Ability to understand and willingness to sign a written informed consent document. • Patient must be accessible to treatment and follow-up procedures
* Fertile women must have a negative pregnancy test. Fertile men and women must use effective contraception. Fertile women included in the study must use effective contraception for the duration of study treatment and one month thereafter.
* Ultra-centrally located tumors are tumors located within the 0.0 to 0.5 cm zone of the trachea, main bronchi or intermediate bronchus. Evaluation is primarily performed on the diagnostic CT scan
* Patients with other non-central tumors synchronous with the central lesion may be included and treated with SBRT in respect to local practice.
* A baseline PET/CT scan within 2 months of inclusion.
* An ablative strategy should be deemed clinically relevant and it is at the discretion of the treating physician to decide.

Exclusion Criteria:

* Tumor with intra-bronchial or intra-tracheal growth, as assessed on a diagnostic CT/MR-scan or endoscopic procedure
* If the patient has received previous radiotherapy, the combined dose at the radiation site must be evaluated by the treating physician and preferably not exceed the dose constraints
* Patient cannot tolerate the physical set up required for SBRT. • Uncontrolled intercurrent illness
* Pregnancy
* Patient participating in another interventional study
* For patients in STAR-LUNG, lack of MR compatibility due to pacemaker, inserted steel or similar.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2033-05-01 (Estimated)

PRIMARY OUTCOMES:
Toxicity: Cumulative CTCAE grade ≥ 4 SABR related toxicity (TRAE) | Assessed at 6 months
  Registration of toxicity will be assessed according to a prespecified selection of organ related adverse events defined by CTCAE version 5.0.
Toxicity: Cumulative CTCAE grade ≥ 4 SABR related toxicity (TRAE) | Assessed at 12 months
  Registration of toxicity will be assessed according to a prespecified selection of organ related adverse events defined by CTCAE version 5.0.
Toxicity: Cumulative CTCAE grade ≥ 4 SABR related toxicity (TRAE) | Assessed at 2 years
  Registration of toxicity will be assessed according to a prespecified selection of organ related adverse events defined by CTCAE version 5.0.
Toxicity: Cumulative CTCAE grade ≥ 4 SABR related toxicity (TRAE) | Assessed at 5 years
  Registration of toxicity will be assessed according to a prespecified selection of organ related adverse events defined by CTCAE version 5.0.

SECONDARY OUTCOMES:
Local progression free survival (LPFS) | Up to 10 years
  Local progression-free survival (LPFS) is defined from the start of radiotherapy treatment until death or date of local recurrence. Events are death and local recurrence.
Overall survival (OS) | Up to 10 years
  Overall survival (OS) is defined as the time from start of radiotherapy treatment until death by any cause.
Disease free survival (DFS) | Up to 10 years
  Disease free survival (DFS) is defined from start of radiotherapy treatment until date of first locoregional or metastatic recurrence or death from any cause. Events are recurrence and death.
Time-to-treatment failure (TTF) | Up to 10 years
  Time-to-treatment failure (TTF) is defined as time from start of radiotherapy treatment until the date of relapse; the patient has withdrawn patient consent or premature termination of SBRT due to toxicity. Events are death due to primary cancer, death due to protocol treatment and date of local, regional or metastatic recurrence.

CONTACTS AND LOCATIONS:
Locations (6):
- Denmark (6):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Herlev University Hospital, Herlev
  - Odense University Hospital, Odense
  - Department of Oncology, Lillebaelt Hospital, Vejle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoffmann L, Persson GF, Nygard L, Nielsen TB, Borrisova S, Gaard-Petersen F, Josipovic M, Khalil AA, Kjeldsen R, Knap MM, Kristiansen C, Moller DS, Ottosson W, Sand H, Thing R, Pohl M, Schytte T. Thorough design and pre-trial quality assurance (QA) decrease dosimetric impact of delineation and dose planning variability in the STRICTLUNG and STARLUNG trials for stereotactic body radiotherapy (SBRT) of central and ultra-central lung tumours. Radiother Oncol. 2022 Jun;171:53-61. doi: 10.1016/j.radonc.2022.04.005. Epub 2022 Apr 11. PMID 35421513